CLINICAL TRIAL: NCT06730555
Title: Project ACCESS: Advancing Access to HIV/HCV Testing Through Transformation in Syringe Services Programs: A Cluster Randomized Trial
Brief Title: Advancing Access to HIV/HCV Testing for People Who Inject Drugs (PWID)
Acronym: ACCESS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Tyler Scott Bartholomew, Associate Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 20240611; R01DA060462 (NIH)
Record Dates: First submitted 2024-12-09; First posted 2024-12-12 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2025-09

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACCESS Group (Experimental): Participants in this group will receive the ACCESS intervention for up to 18 months
  Interventions: Behavioral: ACCESS Intervention
- Control Group (Active Comparator): Participants in this group will receive a link to the CDC Compendium of Evidence-Based Interventions for up to 18 months.
  Interventions: Behavioral: Control Group

INTERVENTIONS:
Behavioral: ACCESS Intervention — Participants will receive the ACCESS intervention with funding, consisting of up to 16 hours of practice facilitation per month in person and/or virtually. Practice facilitation is training and support on implementation of routine HIV/HCV screening.
  Arms: ACCESS Group
Behavioral: Control Group — Participants will receive a link to the CDC compendium of evidence-based interventions for HIV prevention.
  Arms: Control Group

SUMMARY:
The purpose of this study is to test the effectiveness of the ACCESS strategy: an organizational-level intervention that uses funding and practice facilitation to improve the organizational capacity of syringe services programs (SSPs) to implement routine, opt-out HIV and Hepatitis C (HCV) testing and linkage to care for people who inject drugs (PWID).

ELIGIBILITY:
Inclusion Criteria:

* SSPs must:

  1. be operating in an Ending the HIV Epidemic (EHE) or Centers for Disease Control and Prevention (CDC) determined vulnerable jurisdictions;
  2. serve at least 300 unique participants per year;
  3. not currently offer opt-out HIV/HCV testing;
  4. be capable and willing to prospectively collect aggregated, site-level data on the number of participants who are: i) offered HIV/HCV screening, ii) completed these tests, and iii) linked to care, as well as provide participant demographics;
  5. have key staff that consent to participate in study surveys, qualitative interviews and practice facilitation throughout the study.

Exclusion Criteria:

* SSPs must not:

  1. currently receive or have received Frontline Communities in the United States (FOCUS) funding;
  2. have already implemented opt-out HIV/HCV testing.
  3. currently participating in SAIA-SSP-HIV (NCT06025435)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-06-27 (Actual); Primary Completion 2028-08-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Number of SSP participants reached | up to 18 months
  Number of total HIV/HCV tests completed divided by the number of unique individuals seen
Adoption | up to 6 months
  Proportion of SSPs that have created an HIV/HCV opt-out testing policy

SECONDARY OUTCOMES:
Number of SSP participants reached after the intervention | up to 30 months
  Number of total HIV/HCV tests completed divided by the number of unique individuals seen

CONTACTS AND LOCATIONS:
Overall Officials: Tyler Bartholomew, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No